CLINICAL TRIAL: NCT05903066
Title: TRansmural hEaliNg Definition in CroHn's Disease - The TRENCH1 Study
Brief Title: TRansmural hEaliNg Definition in CroHn's Disease (TRENCH 1)
Acronym: TRENCH 1
Status: Recruiting | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID-2022-03
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Crohn Disease
Keywords: IBD; CD
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, stool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Magnetic Resonance Enterography (MRE) — MRE performed as part of the standard of care follow up of the patient, the exam will be recorded for the study and analysed by central readers.

SUMMARY:
Multicenter prospective cross-sectional study of CD patients, its aim is the construction of an objective and reproducible system for evaluation of Transmural healing in Crohn's Disease (CD).

Primary objective : Objective definition of depth or grade of transmural healing in relation to radiologic signs observed during Magnetic Resonance Enterography (MRE) in CD

DETAILED DESCRIPTION:
Number of patients : 210 patients, in 14 sites (only one investigator per site), 15 patients per site, 5 patients per grade of transmural healing based on the appraisal of a local reader pair (a gastroenterologist and a radiologist).

Recruitment period : 2 years

Primary Endpoint : Objective definition of depth or grade of transmural healing in relation to radiologic signs observed during Magnetic Resonance Enterography (MRE) in CD

Secondary Endpoints :

* To analyze intra- and inter-observer variability of radiological findings.
* To analyze intra- and inter-observer variability of TH definitions in CD.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Patient diagnosed with CD for more than 6 months with histological confirmation available in his medical record.
* Indication for MRE based on routine clinical practice validated by the treating physician
* Any CD treatment will be authorized, such as biologicals (infliximab, adalimumab, vedolizumab, ustekinumab…), or immunomodulators (azathioprine, 6-mercaptopurine, methotrexate…).
* The subjects sign and date a written, informed consent form and any required privacy authorization prior to the initiation of the study.
* A subject can be enrolled into the study only if the grade of TH (assessed by the LRP) corresponding to the subject is not already fulfilled.

Exclusion Criteria:

* Pregnancy during the study
* People unable to give consent (because of their physical or mental state)
* Absence of written consent
* Ulcerative colitis or unclassified IBD
* Specific postsurgical settings: ileoanal anastomosis, ileostomy or colostomy.
* Less than 3 evaluable ileocolic segments or more than 3 resected ileocolonic segments (not counting ileocecal valve)
* Severe obstructive symptoms
* Symptomatic intra-abdominal abscess
* Contraindication for MRI
* Isolated perianal disease without luminal location
* MRE images of poor quality, based on previously defined criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CD for more than 6 months with histological confirmation available in his medical record, with an indication for MRE based on routine clinical practice validated by the treating physician
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Objective definition of depth or grade of transmural healing in relation to radiologic signs observed during Magnetic Resonance Enterography (MRE) in CD | Day 1
  An index (depth of remission) or score (grade of remission) will be constructed through multiple linear or logistic mixed regression models.

SECONDARY OUTCOMES:
Intra- and inter-observer variability of lesions observed per segment during MRE in CD | Day 1
  Variations in MRE readings images between the CR will be quantified through the Kappa coefficient for qualitative items and through the intraclass correlation coefficient for quantitative items.
Intra- and inter-observer variability of depth and grade of global transmural healing in CD | Day 1
  Variations in MRE readings images between the CR will be quantified through the Kappa coefficient for qualitative items and through the intraclass correlation coefficient for quantitative items.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie GEYL, Principal Investigator — CHU Limoge Dupuytren
Locations (18):
- CHU de Liège, Liège, Belgium
- France (17):
  - CHU Amiens-Picardie (site Sud), Amiens
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Bordeaux
  - APHP - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Clermont-Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - APHP - Hôpital Louis Mourier, Colombes
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU Limoges Dupuytren, Limoges
  - AP-HM - Hôpital Nord, Marseille
  - CHU de Montpellier - Hôpital Saint Eloi, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice - Hôpital l'Archet II, Nice
  - CHU de Nîmes - Hôpital Carémeau, Nîmes
  - APHP - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - CHRU de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy